CLINICAL TRIAL: NCT02255682
Title: Living With Statins - The Impact of Cholesterol Lowering Drugs on Health, Lifestyle and Well-being
Acronym: LIFESTAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Flemming Dela, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: LIFESTAT - Observational Study
Record Dates: First submitted 2014-09-12; First posted 2014-10-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Cardiovascular Disease; Diabetes Mellitus
Keywords: physical activity; statin therapy; diabetes mellitus; cardiovascular disease; Q10-supplementation
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Motor Activity | interventions — Simvastatin; Tuberculin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin and Q10-placebo (Placebo Comparator): Simvastatin 40 mg orally administered daily and Q10-placebo for 8 weeks
  Interventions: Drug: Simvastatin
- Simvastatin and Q10 (Active Comparator): Simvastatin 40 mg orally administered daily for 8 weeks in combination with Q10 supplementation of 400 mg/daily
  Interventions: Drug: Simvastatin; Dietary Supplement: Q10

INTERVENTIONS:
Drug: Simvastatin
  Other Names: Simvastatin Actavis; Simvastatin Hexal; Simvastatin KRKA; Simvastatin Orion; Simvastatin Sandoz; Simvastatin Stada; Simvastatin Teva; Zocor
Dietary Supplement: Q10
  Other Names: Bioquinon Q10
  Arms: Simvastatin and Q10

SUMMARY:
Background Statins are cholesterol lowering drugs that are prescribed to lower the risk of cardio-vascular diseases. The use of statins has increased markedly and it is now one of the most prescribed drugs in the world. 600,000 people in Denmark are taking statins on a daily basis, 40 % of these are taking the medication without having any other risk factors for cardio-vascular diseases than elevated blood-cholesterol i.e. they are in primary prevention.

Statins are not without side effects and studies have shown that there is an elevated risk of developing diabetes when taking statins. This has led to an increased debate about the use of statins in primary prevention. Furthermore a large meta-analysis has shown that to prevent one event of cardio-vascular disease, it is necessary to treat 200 people for 3-5 years. These data suggest that more conservative use of statins to prevent CVD in otherwise healthy individuals at low risk for future CVD may be warranted.

Other side effects of statins are muscle myalgia, muscle cramps and fatigue which potentially can prevent a physically active lifestyle. The biomedical background of these side effects is not fully elucidated but it has been shown that there is a link to decreasing levels of an important enzyme, Q10, which plays a role in muscle energy metabolism.

Hypothesis

The overarching research question is: why does statin treatment cause muscle pain? Does statin treatment impair (or even prevent) physical exercise training? Furthermore we would like to answer the following questions:

1. Does statin treatment impair (or even prohibit) physical exercise training?
2. Does statin treatment cause:

   * Decreased muscle strength?
   * Skeletal muscle inflammation?
   * Decreased mitochondrial respiratory function?
3. Abnormal glucose homeostasis?

DETAILED DESCRIPTION:
Background

HYPERCHOLESTEROLEMIA AND STATIN USE IN DENMARK

Simvastatin is the most commonly prescribed statin, a class of drugs that inhibit hydroxyl-methyl-glutaryl (HMG) coenzyme A reductase, and thereby blocking biosynthesis of cholesterol in the liver. Simvastatin is prescribed for individuals with elevated low-density lipoprotein cholesterol (LDL-C) and/or total cholesterol, because these clinical parameters are viewed as a risk factor for cardiovascular-disease (CVD), even in the absence of other health problems or risk factors, such as previous myocardial infarction, diabetes or hypertension.

Approximately 40% of the prescriptions for statins are issued for primary prevention of elevated cholesterol by general practitioners to patients without bodily symptoms or signs. Only the "cholesterol number" makes the risk of heart attack and stroke visible. The lack of symptoms is likely to be of importance for patients' adherence to treatment as is adverse effects. A number of factors, such as information in mass media and changes in daily life, may affect the decision to take the treatment

TREATMENT GUIDELINES FOR HYPERCHOLESTEROLEMIA

The guidelines (8; 10) indicate preventive treatment with statins is appropriate in individuals with >10% predicted risk of a major vascular event within 5 years, while, some, but not all opinion-leaders advocate a 5% threshold (2; 8). Nevertheless, statin therapy failed to reduce all-cause mortality in a meta-study of 65,229 patients without CVD, some of whom had diabetes (11). Similarly, a Cochrane review analysis, which included some studies in which more than 10% of the patients had history of CVD, showed only 0.5% reduction in all-cause mortality, indicating that for every 200 patients taking statins daily for 5 years, 1 death would be prevented (13). These data suggest that more conservative use of statins to prevent CVD in otherwise healthy individuals at low risk for future CVD may be warranted.

THE DOWN-SIDE

Rhabdomyolysis (skeletal muscle cell death) is an infrequent but serious side-effect of statin use, that can on rare occasion lead to acute renal failure and death (i.e., 1.5 deaths per 106 prescriptions (9)). Statin use is much more frequently associated with muscle dysfunction, including myalgia (muscle pain), cramps, and weakness. The reported incidence of myalgia varies from 1% (pharmaceutical company reports) to as high as 75% in statin-treated athletes (7; 9). Mild to severe myalgia is a strong disincentive to regular exercise, and because regular exercise is one of the critical life-style approaches to preventing CVD and reducing blood cholesterol, this is a significant down-side of statin use. Regular exercise is also effective in preventing and treating obesity and type 2 diabetes, which themselves are risk factors for CVD (16).

The mechanism behind the myalgia is not known. However, we have recently demonstrated that muscle mitochondrial function is impaired with statin treatment and the Q10 protein may play a key role in this (6). In addition, the statins also negatively affect the glucose tolerance (6), increasing the risk of type 2 diabetes.

RESEARCH QUESTIONS:

The overarching research question is: why does statin treatment cause muscle pain? We are not the only research group in the world that try to answer that question, but we are the only one that has indeed provided a mechanistic explanation, and provided a proof-of-concept (6). We will now test this in a larger patient population.

Our background in muscle and exercise physiology and in bioenergetics makes it natural to further ask:

1. Does statin treatment impair (or even prohibit) physical exercise training?
2. Does statin treatment cause:

   * Decreased muscle strength?
   * Skeletal muscle inflammation?
   * Decreased mitochondrial respiratory function?
3. Abnormal glucose homeostasis?

Re question B & C: If so, can physical training counteract this effect of statin treatment?

Methodology

COHORT

Patients that fulfil defined inclusion and exclusion criteria will be recruited from General Practice clinics in Copenhagen and news paper advertisements. The vast majority of these patients are being treated on basis of the HeartScore risk estimation system that offers direct estimation of the ten-year risk of fatal cardiovascular disease in a format suited to the constraints of clinical practice (14) (www.HeartScore.org).

60 patients both men and women (age: 40-70 years; BMI: 25-35 kg/m2) taking Simvastatin as primary prevention are recruited. No other risk factors for CVD except elevated total cholesterol and/or elevated LDL cholesterol and mild hypertension (<145/100 mm Hg) must be present.

The patients will be allocated (randomization by drawing a lot) to one of two groups:

* Simvastatin 40 mg/day and Q10-supplementation 400 mg/day
* Simvastatin 40 mg/day and Q10-placebo The intervention period is 8 weeks with a series of experimental days before and after.

Experimental days (identical before and after the interventions):

Day 1 (½ day - overnight fasting):

* Medical history; clinical examination + ECG. Measurements: Blood pressure, weight, height, W/H-ratio, thigh circumference.
* Dual Energy X-ray Absorptiometry-scan (DXA) (body composition and body fat).
* FatMax test and maximal oxygen uptake test (VO2-max) or ergometer bike.

Day 2 (½ day - overnight fasting):

* Oral glucose tolerance test + score questionnaire for muscle pain/discomfort (Visual Analog Scale) and a questionnaire regarding the extent of muscle pain/discomfort.
* Isokinetic strength and Rate of Force Development (PowerRig and KinCom dynamometer).
* Repeated VO2-max-test

Day 3 (1 day - overnight fasting):

* Muscle biopsy, vastus lateralis (before and after clamp), fat biopsy from subcutaneus adipose tissue in the abdomen.
* Intravenous glucose tolerance test (IVGTT)
* Euglycemic, hyperinsulinaemic clamp.

Statistical considerations

The major end-points are all end-point which we have tested before in other clinical populations. In general, in order to detect a 10% difference in these parameters before vs. after a training program or between statin users and control, requires 15-20 subjects in each group if an alpha level of <0.05 and risk of type 2 error is set to 10%. 10-15 subjects are necessary if the "conventional" 20% type 2 error risk is implemented. Thus, the present study has a considerable safety-margin in terms of statistical power.

ELIGIBILITY:
Inclusion Criteria:

* 40-70 years.
* BMI 25-35.
* prescribed Simvastatin 40 mg/daily by their general practitioner.

Exclusion Criteria:

* Diabetes Mellitus.
* Cardiovascular disease such as arrythmia, ischaemic heart disease.
* Musculoskeletal disorders preventing the subject to perform physical.
* Mental disorders preventing the subject to understand the project description.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Difference in myalgia | 8 weeks
  Difference in myalgia, measured by visual analog scale (VAS) between Simvastatin treated patients receiving Q10 or Q10-placebo.

SECONDARY OUTCOMES:
Difference in VO2-max | 8 weeks
  Difference in VO2-max in Simvastatin treated patients receiving Q10 or Q10-placebo.
Difference in muscle strength | 8 weeks
  Difference in muscle strength in Simvastatin treated patients receiving Q10 or Q10-placebo.
Difference in glucose metabolism | 8 weeks
  Difference in glucose metabolism in Simvastatin treated patients receiving Q10 or Q10-placebo.
Difference in mitochondrial function | 8 weeks
  Difference in mitochondrial function in Simvastatin treated patients receiving Q10 or Q10-placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, MD, MDSci, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boushel R, Gnaiger E, Schjerling P, Skovbro M, Kraunsoe R, Dela F. Patients with type 2 diabetes have normal mitochondrial function in skeletal muscle. Diabetologia. 2007 Apr;50(4):790-6. doi: 10.1007/s00125-007-0594-3. Epub 2007 Feb 15. PMID 17334651
- [Background] Ebrahim S, Casas JP. Statins for all by the age of 50 years? Lancet. 2012 Aug 11;380(9841):545-7. doi: 10.1016/S0140-6736(12)60694-1. Epub 2012 May 17. No abstract available. PMID 22607823
- [Background] Larsen S, Hey-Mogensen M, Rabol R, Stride N, Helge JW, Dela F. The influence of age and aerobic fitness: effects on mitochondrial respiration in skeletal muscle. Acta Physiol (Oxf). 2012 Jul;205(3):423-32. doi: 10.1111/j.1748-1716.2012.02408.x. Epub 2012 Feb 11. PMID 22212519
- [Background] Larsen S, Nielsen J, Hansen CN, Nielsen LB, Wibrand F, Stride N, Schroder HD, Boushel R, Helge JW, Dela F, Hey-Mogensen M. Biomarkers of mitochondrial content in skeletal muscle of healthy young human subjects. J Physiol. 2012 Jul 15;590(14):3349-60. doi: 10.1113/jphysiol.2012.230185. Epub 2012 May 14. PMID 22586215
- [Background] Larsen S, Stride N, Hey-Mogensen M, Hansen CN, Andersen JL, Madsbad S, Worm D, Helge JW, Dela F. Increased mitochondrial substrate sensitivity in skeletal muscle of patients with type 2 diabetes. Diabetologia. 2011 Jun;54(6):1427-36. doi: 10.1007/s00125-011-2098-4. Epub 2011 Mar 18. PMID 21424396
- [Background] Larsen S, Stride N, Hey-Mogensen M, Hansen CN, Bang LE, Bundgaard H, Nielsen LB, Helge JW, Dela F. Simvastatin effects on skeletal muscle: relation to decreased mitochondrial function and glucose intolerance. J Am Coll Cardiol. 2013 Jan 8;61(1):44-53. doi: 10.1016/j.jacc.2012.09.036. PMID 23287371
- [Background] Singh P, Kohr D, Kaps M, Blaes F. Skeletal muscle cell MHC I expression: implications for statin-induced myopathy. Muscle Nerve. 2010 Feb;41(2):179-84. doi: 10.1002/mus.21479. PMID 19813190
- [Background] Cholesterol Treatment Trialists' (CTT) Collaborators; Mihaylova B, Emberson J, Blackwell L, Keech A, Simes J, Barnes EH, Voysey M, Gray A, Collins R, Baigent C. The effects of lowering LDL cholesterol with statin therapy in people at low risk of vascular disease: meta-analysis of individual data from 27 randomised trials. Lancet. 2012 Aug 11;380(9841):581-90. doi: 10.1016/S0140-6736(12)60367-5. Epub 2012 May 17. PMID 22607822
- [Background] Parker BA, Thompson PD. Effect of statins on skeletal muscle: exercise, myopathy, and muscle outcomes. Exerc Sport Sci Rev. 2012 Oct;40(4):188-94. doi: 10.1097/JES.0b013e31826c169e. PMID 23000957
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren WM, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte Op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; Comitato per Linee Guida Pratiche (CPG) dell'ESC. [European Guidelines on Cardiovascular Disease Prevention in Clinical Practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and other societies on cardiovascular disease prevention in clinical practice (constituted by representatives of nine societies and by invited experts)]. G Ital Cardiol (Rome). 2013 May;14(5):328-92. doi: 10.1714/1264.13964. No abstract available. Italian. PMID 23612326
- [Background] Ray KK, Seshasai SR, Erqou S, Sever P, Jukema JW, Ford I, Sattar N. Statins and all-cause mortality in high-risk primary prevention: a meta-analysis of 11 randomized controlled trials involving 65,229 participants. Arch Intern Med. 2010 Jun 28;170(12):1024-31. doi: 10.1001/archinternmed.2010.182. PMID 20585067
- [Background] Ridker PM, Pradhan A, MacFadyen JG, Libby P, Glynn RJ. Cardiovascular benefits and diabetes risks of statin therapy in primary prevention: an analysis from the JUPITER trial. Lancet. 2012 Aug 11;380(9841):565-71. doi: 10.1016/S0140-6736(12)61190-8. PMID 22883507
- [Background] Taylor F, Ward K, Moore TH, Burke M, Davey Smith G, Casas JP, Ebrahim S. Statins for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD004816. doi: 10.1002/14651858.CD004816.pub4. PMID 21249663
- [Derived] Dohlmann TL, Morville T, Kuhlman AB, Chrois KM, Helge JW, Dela F, Larsen S. Statin Treatment Decreases Mitochondrial Respiration But Muscle Coenzyme Q10 Levels Are Unaltered: The LIFESTAT Study. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2501-2508. doi: 10.1210/jc.2018-01185. PMID 30299473